CLINICAL TRIAL: NCT00659763
Title: Diagnostic Strategies in Patients Suspected of Irritable Bowel Syndrome and the Prevalence of Intestinal Parasites in Patients Suspected of Irritable Bowel Syndrome
Brief Title: Diagnostic Strategies in Patients Suspected of Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Statens Serum Institut (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Line Oestergaard Engsbro, MD, phD-student, Zealand University Hospital
Other Study IDs: SJ-40
Record Dates: First submitted 2008-04-03; First posted 2008-04-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Diagnosis
MeSH Terms: conditions — Irritable Bowel Syndrome; Disease | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and fecal sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients suspected of irritable bowel syndrome referred from GP´s, who fulfill the ROM III criteria for IBS
  Interventions: Other: Exclusion diagnosis
- B: Patients suspected of irritable bowel syndrome referred from GP´s, who fulfill he ROME III criteria for IBS
  Interventions: Other: Clinical diagnosis

INTERVENTIONS:
Other: Exclusion diagnosis — Patient fulfill ROME III criteria No Alarmsignals Blood tests: FBC,CRP, ALAT, bilirubins, bas.phosphatases, Albumine, TSH, calcium, celiac screening, lactase gene test.
  3 consecutive fecal samples for worm, ovaes and parasites Sigmoidoscopy with biopsy
  Groups: A
Other: Clinical diagnosis — Patient fulfill ROME III criteria No Alarm signals Blood tests: FBC, CRP.
  Groups: B

SUMMARY:
The purpose of this study is to determine whether a clinical diagnosis of irritable bowel syndrome based on patient reported symptoms and a few blood tests is safe, and to determine whether a clinical diagnosis is as good for the patient and as economical for the society as a diagnosis based on exclusion of a number of organic diseases by performing a number of blood tests, fecal analyzes and a scopic examination of bowel.

The purpose of the second part of the study is to determine which intestinal parasites the patients have in their bowel and whether these parasites are the cause of the disease.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* consultant in general practice for gastrointestinal symptoms, where the GP suspects irritable bowel syndrome
* full fill the ROME III criteria
* signed informed consent

Exclusion Criteria:

* alarm signals
* pregnancy
* comorbid diseases, that interfere with primary endpoint
* medicine and alcohol abuse
* patient do not speak or understand danish
* investigations for irritable bowel syndrome with in the last 3 years

from november 2008: patients aged above 40 with a duration shorter than one year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are recruited from primary care.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
health related quality of life measured by SF-36 | baseline and after 1 year

SECONDARY OUTCOMES:
Symptoms measured by GSRS and GSRS-IBS | baseline, every month for a year and after 1 year
sick days and reduced productivity measured by WPAI:IBS | baseline, every month and after 1 year
differential diagnoses in both arms | 1 year
Health related quality of life measured by IBS-QOL measurement | baseline and after 1 year
The overall satisfaction with the diagnostic strategy | after initial diagnostic work up and after 1 year
The use of resources in the health care system measured by the number of doctor visits, ambulatory visits, emergency room visits, hospitalizations and diagnostic tests over 1 year follow up. | every month and after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Line OE Engsbro, MD, Principal Investigator — Køge Hospital; Peter Bytzer, Professor MD, Study Chair — Køge Hospital
Locations (1):
- Medical Departement, Koege Hospital, Køge, Denmark

REFERENCES:
- [Derived] Engsbro AL, Begtrup LM, Haastrup P, Storsveen MM, Bytzer P, Kjeldsen J, Schaffalitzky De Muckadell O, Jarbol DE. A positive diagnostic strategy is safe and saves endoscopies in patients with irritable bowel syndrome: A five-year follow-up of a randomized controlled trial. Neurogastroenterol Motil. 2021 Mar;33(3):e14004. doi: 10.1111/nmo.14004. Epub 2020 Oct 7. PMID 33029843
- [Derived] Larsen AR, Engsbro AL, Bytzer P. Screening instruments for anxiety and depression in patients with irritable bowel syndrome are ambiguous. Dan Med J. 2014 Feb;61(2):A4785. PMID 24495890
- [Derived] Begtrup LM, Engsbro AL, Kjeldsen J, Larsen PV, Schaffalitzky de Muckadell O, Bytzer P, Jarbol DE. A positive diagnostic strategy is noninferior to a strategy of exclusion for patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Aug;11(8):956-62.e1. doi: 10.1016/j.cgh.2012.12.038. Epub 2013 Jan 26. PMID 23357491